CLINICAL TRIAL: NCT05535400
Title: Effects of a Physical-Psychological Integrative (PPI) Intervention on Physical Inactivity, Depression and Chronic Pain for Community-Dwelling Spinal Cord Injury Survivors: a Pilot Randomized Controlled Trial
Brief Title: Effects of Physical-Psychological Integrative Intervention on SCI Patient: a Pilot Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P0038951
Record Dates: First submitted 2022-07-11; First posted 2022-09-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2022-06

CONDITIONS: Spinal Cord Injuries; Physical Inactivity; Depression; Chronic Pain
Keywords: Spinal cord injuries; Physical Psychological Integrative
MeSH Terms: conditions — Spinal Cord Injuries; Sedentary Behavior; Depression; Chronic Pain

STUDY DESIGN:
Intervention Model Description: We aim to have two study group, including the eight-week Physical-Psychological Integrative online intervention group and the brief online didactic education control group.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The participants could not be blinded due to the nature of the intervention. Patients will be reminded to keep the intervention content confidential and not discuss this with participants in the control group to avoid contamination. Also, the research assistant (RA1) who responsible for assessing all the outcomes will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Physical-Psychological Integrative (PPI) intervention group (Experimental): The PPI intervention will include eight weekly online group sessions (with each session lasts for 60-90 minutes). At the beginning of each online group meeting, the intervention provider will use motivational interviewing techniques to promote participants' adherence to the physical activity program, followed by on-line group psychological intervention
  Interventions: Behavioral: Physical-Psychological Integrative Intervention
- The brief online didactic education control group (Active Comparator): Participants in the control group will receive a short video call (approximately 20 minutes each week for eight weeks) from the trained research assistant, i.e., RA 2 to provide general physical and psychological suggestions (e.g., encouragement of performing physical activities, and communication skills with family members/friends, and engagement in the community life). This is to control the contact effects of the PPI intervention.
  Interventions: Device: Brief online didactic education

INTERVENTIONS:
Behavioral: Physical-Psychological Integrative Intervention — The PPI intervention will include eight weekly online group sessions (with each session lasts for 60-90 minutes). At the beginning of each online group meeting, the intervention provider will use motivational interviewing techniques to promote participants' adherence to the physical activity program. And the content of the intervention includes eight different sessions, including Session 1- Orientation and engagement, Session 2- Awareness and Acceptance; Session 3- Non-judgement; Session 4- Stay present and let go; Session 5- Our thoughts are not real & Response without reacting; Session 6- Empowerment of self-management and discuss pain management; Session 7- Seek out pleasant things and social support and Session 8- Review the intervention and end the programme.
  Arms: The Physical-Psychological Integrative (PPI) intervention group
Device: Brief online didactic education — Participants in the control group will receive a short video call (approximately 20 minutes each week for eight weeks) from the trained research assistant, i.e., RA 2 to provide general physical and psychological suggestions (e.g., encouragement of performing physical activities, and communication skills with family members/friends, and engagement in the community life). This is to control the contact effects of the PPI intervention.
  Arms: The brief online didactic education control group

SUMMARY:
Spinal cord injury (SCI) is a neurological disorder that leads to "partial or complete loss of people's motor and/ or sensory function below the level of the injury".

The PPI intervention group participants will indicate significantly greater improvements when compared with those in control group in the minutes of performing the moderate-to-rigorous physical activity, depression, chronic pain and mindfulness skills and quality of life at post-intervention, and three months follow-up. The use of psychological motivational interviewing and online face-to-face meetings will be good modalities for the people with SCI to overcome the barriers of not having face-to-face interactions and transportation problems. And the intervention would be feasible and improve SCI people's physical inactivity, depression and chronic pain as to step up the control of the modifiable risk factors for non-communicable diseases.

DETAILED DESCRIPTION:
This study is a two-arm, single-blind pilot randomized controlled trial, and it will be adopted to evaluate or compare the effects between the Physical-Psychological Integrative (PPI) intervention group and the brief online didactic education control group.

Seventy-two participants will be recruited from the Hong Kong Direction Association for the Handicapped. 36 people with SCI will be assigned to intervention or control group. Participants in PPI Intervention group will receive a Fitbug wristband activity trackers and exercise bands as an incentive and encouragement for doing more physical exercises. The intervention includes eight weekly online group sessions. Qualitative interviews with the PPI intervention group participants will be conducted to understand their acceptance and perceived strengths and limitations of the intervention programme. While the one in the control group will receive a short video call for general physical and psychological suggestions. This can help to control the contact effects of the PPI intervention. Primary outcomes will be leisure-time physical activity, depression and chronic pain. Secondary outcome will be exercise efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years older;
* Currently living in the community and having SCI for more than 6 months;
* Complete injury at the C6 or below or incomplete injury at any level ;
* Having a computer/ smartphone with audio-speaking function and Zoom software, and internet access in a secure place;
* Using a wheelchair for at least 2 hours a day and having the approval from the physicians to perform exercises;
* Having no problems in hearing, verbal communication, and vision;
* Able to communicate in Cantonese and to provide informed consent.

Exclusion Criteria:

* Presented with any significant cognitive impairment or brain injury;
* Engaged in ongoing psychotherapy or any other physiotherapy/ exercise/ relaxation interventions;
* Physically active for more than 150 minutes per week;
* Experiencing significant psychotic symptoms, substance misuse or medically not able for the exercise and psychological programme as diagnosed by their physicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Leisure-time Physical Activity | Leisure-time Physical Activity will be assessed throughout the study period, an average of two months.
  Participants' leisure-time moderated-to-rigorous physical activity (MVPA) will be assessed by using the Fitbug Orb (Chicago, IL) which is a wearable, display, triaxial accelerometer that pairs with Bluetooth with compatible smartphones.
Depression at post-test | Depression will be assessed at post-intervention, an average of two months.
  The 9-item Patient Health Questionnaire (PHQ-9) will be used to measure the participants' depression level.
Depression at three months follow-up | Depression will be assessed after three months follow-up.
  The 9-item Patient Health Questionnaire (PHQ-9) will be used to measure the participants' depression level.
Chronic pain at post test | Chronic pain will be assessed at post-intervention, an average of two months.
  An 11-point numerical pain rating scale (NPRS) will be used to measure pain intensity and pain unpleasantness (in the past week), where zero means no pain and 10 means the worst imaginable pain.
Chronic pain at three months follow-up | Chronic pain will be assessed after three months follow-up.
  An 11-point numerical pain rating scale (NPRS) will be used to measure pain intensity and pain unpleasantness (in the past week), where zero means no pain and 10 means the worst imaginable pain.

SECONDARY OUTCOMES:
Exercise Efficacy at post test | Exercise efficacy will be assessed at post-intervention, an average of two months.
  A scale aim at testing people's confidence to continue exercising in the face of barriers to exercise.
Exercise Efficacy at three months follow-up | Exercise Efficacy will be assessed after three months follow-up.
  A scale aim at testing people's confidence to continue exercising in the face of barriers to exercise.
Mindfulness at post test | Mindfulness will be assessed at post-intervention, an average of two months.
  The 39-item Five Facet Mindfulness Questionnaire (FFMQ) will be used to measuring the five aspects of mindfulness including observing, describing, acting with awareness, non-judgmental and non-reactive.
Mindfulness at three months follow-up | Mindfulness will be assessed after three months follow-up.
  The 39-item Five Facet Mindfulness Questionnaire (FFMQ) will be used to measuring the five aspects of mindfulness including observing, describing, acting with awareness, non-judgmental and non-reactive.
QoL: Quality of Life at post test | Quality of Life will be assessed at post-intervention, an average of two months.
  The 26-item World Health Organization Quality of Life Brief Scale will be used for assessing participants' quality of life.
QoL: Quality of Life at three months follow up | Quality of Life will be assessed after three months follow-up.
  The 26-item World Health Organization Quality of Life Brief Scale will be used for assessing participants' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Dr, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic Unviersity, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alizadeh A, Dyck SM, Karimi-Abdolrezaee S. Traumatic Spinal Cord Injury: An Overview of Pathophysiology, Models and Acute Injury Mechanisms. Front Neurol. 2019 Mar 22;10:282. doi: 10.3389/fneur.2019.00282. eCollection 2019. PMID 30967837
- [Background] March ICfCoSCIPJI. Global summary of spinal cord injury, incidence and economic impact. 2004.
- [Background] Margolis JM, Juneau P, Sadosky A, Cappelleri JC, Bryce TN, Nieshoff EC. Health care resource utilization and medical costs of spinal cord injury with neuropathic pain in a commercially insured population in the United States. Arch Phys Med Rehabil. 2014 Dec;95(12):2279-87. doi: 10.1016/j.apmr.2014.07.416. Epub 2014 Aug 24. PMID 25159715
- [Background] Hu Y, Mak JN, Wong YW, Leong JC, Luk KD. Quality of life of traumatic spinal cord injured patients in Hong Kong. J Rehabil Med. 2008 Feb;40(2):126-31. doi: 10.2340/16501977-0150. PMID 18509577
- [Background] Martin Ginis KA, Jetha A, Mack DE, Hetz S. Physical activity and subjective well-being among people with spinal cord injury: a meta-analysis. Spinal Cord. 2010 Jan;48(1):65-72. doi: 10.1038/sc.2009.87. Epub 2009 Jul 7. PMID 19581918
- [Background] Quel de Oliveira C, Refshauge K, Middleton J, de Jong L, Davis GM. Effects of Activity-Based Therapy Interventions on Mobility, Independence, and Quality of Life for People with Spinal Cord Injuries: A Systematic Review and Meta-Analysis. J Neurotrauma. 2017 May 1;34(9):1726-1743. doi: 10.1089/neu.2016.4558. Epub 2016 Dec 20. PMID 27809702
- [Background] Khazaeipour Z, Taheri-Otaghsara SM, Naghdi M. Depression Following Spinal Cord Injury: Its Relationship to Demographic and Socioeconomic Indicators. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):149-55. doi: 10.1310/sci2102-149. Epub 2015 Apr 12. PMID 26364284
- [Background] Bombardier CH, Richards JS, Krause JS, Tulsky D, Tate DG. Symptoms of major depression in people with spinal cord injury: implications for screening. Arch Phys Med Rehabil. 2004 Nov;85(11):1749-56. doi: 10.1016/j.apmr.2004.07.348. PMID 15520969
- [Background] Hadjipavlou G, Cortese AM, Ramaswamy B. Spinal cord injury and chronic pain. BJA Education. 2016;16(8):264-8.
- [Background] Avluk OC, Gurcay E, Gurcay AG, Karaahmet OZ, Tamkan U, Cakci A. Effects of chronic pain on function, depression, and sleep among patients with traumatic spinal cord injury. Ann Saudi Med. 2014 May-Jun;34(3):211-6. doi: 10.5144/0256-4947.2014.211. PMID 25266180
- [Background] Best KL, Routhier F, Sweet SN, Lacroix E, Arbour-Nicitopoulos KP, Borisoff JF. Smartphone-Delivered Peer Physical Activity Counseling Program for Individuals With Spinal Cord Injury: Protocol for Development and Pilot Evaluation. JMIR Res Protoc. 2019 Mar 22;8(3):e10798. doi: 10.2196/10798. PMID 30901001
- [Background] Bombardier CH, Dyer JR, Burns P, Crane DA, Takahashi MM, Barber J, Nash MS. A tele-health intervention to increase physical fitness in people with spinal cord injury and cardiometabolic disease or risk factors: a pilot randomized controlled trial. Spinal Cord. 2021 Jan;59(1):63-73. doi: 10.1038/s41393-020-0523-6. Epub 2020 Jul 21. PMID 32694748
- [Background] Boldt I, Eriks-Hoogland I, Brinkhof MW, de Bie R, Joggi D, von Elm E. Non-pharmacological interventions for chronic pain in people with spinal cord injury. Cochrane Database Syst Rev. 2014 Nov 28;2014(11):CD009177. doi: 10.1002/14651858.CD009177.pub2. PMID 25432061
- [Background] Fann JR, Crane DA, Graves DE, Kalpakjian CZ, Tate DG, Bombardier CH. Depression treatment preferences after acute traumatic spinal cord injury. Arch Phys Med Rehabil. 2013 Dec;94(12):2389-2395. doi: 10.1016/j.apmr.2013.07.004. Epub 2013 Jul 16. PMID 23872078
- [Background] Heutink M, Post MW, Luthart P, Schuitemaker M, Slangen S, Sweers J, Vlemmix L, Lindeman E. Long-term outcomes of a multidisciplinary cognitive behavioural programme for coping with chronic neuropathic spinal cord injury pain. J Rehabil Med. 2014 Jun;46(6):540-5. doi: 10.2340/16501977-1798. PMID 24818861
- [Background] Hearn JH, Finlay KA. Internet-delivered mindfulness for people with depression and chronic pain following spinal cord injury: a randomized, controlled feasibility trial. Spinal Cord. 2018 Aug;56(8):750-761. doi: 10.1038/s41393-018-0090-2. Epub 2018 Mar 26. PMID 29581519
- [Background] Hearn JH, Cross A. Mindfulness for pain, depression, anxiety, and quality of life in people with spinal cord injury: a systematic review. BMC Neurol. 2020 Jan 21;20(1):32. doi: 10.1186/s12883-020-1619-5. PMID 31964353
- [Background] Vall J, Costa CM, Pereira LF, Friesen TT. Application of International Classification of Functioning, Disability and Health (ICF) in individuals with spinal cord injury. Arq Neuropsiquiatr. 2011 Jun;69(3):513-8. doi: 10.1590/s0004-282x2011000400020. PMID 21755132
- [Background] Li Y, Chien WT, Bressington D. Effects of a coping-oriented supportive programme for people with spinal cord injury during inpatient rehabilitation: a quasi-experimental study. Spinal Cord. 2020 Jan;58(1):58-69. doi: 10.1038/s41393-019-0320-2. Epub 2019 Jun 28. PMID 31253849
- [Background] Li Y, Bressington D, Chien WT. Pilot evaluation of a coping-oriented supportive program for people with spinal cord injury during inpatient rehabilitation. Disabil Rehabil. 2019 Jan;41(2):182-190. doi: 10.1080/09638288.2017.1386238. Epub 2017 Oct 10. PMID 28994618
- [Background] Strategy and Action Plan to Prevent and Control Non-communicable Diseases in Hong Kong. Food and Health Burean, Hong Kong.
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Richardson L. Motivational interviewing: helping patients move toward change. J Christ Nurs. 2012 Jan-Mar;29(1):18-24; quiz 25-6. doi: 10.1097/cnj.0b013e318238e510. PMID 22359830
- [Background] Burch V, Penman D. Mindfulness for health: a practical guide to relieving pain, reducing stress and restoring wellbeing: Hachette UK; 2013.
- [Background] Veerubhotla A, Hong E, Knezevic S, Spungen A, Ding D. Estimation of Physical Activity Intensity in Spinal Cord Injury Using a Wrist-Worn ActiGraph Monitor. Arch Phys Med Rehabil. 2020 Sep;101(9):1563-1569. doi: 10.1016/j.apmr.2020.05.014. Epub 2020 Jun 2. PMID 32502566
- [Derived] Li Y, Li M, Bressington D, Li K, Wong AY, Chung WM, Molassiotis A, Ma CZ, Kor PPK, Yeung WF. Effect of a Mindfulness and Motivational Interviewing-Oriented Physical-Psychological Integrative Intervention for Community-Dwelling Spinal Cord Injury Survivors: A Mixed-Methods Randomized Controlled Trial. Arch Phys Med Rehabil. 2024 Sep;105(9):1632-1641. doi: 10.1016/j.apmr.2024.05.017. Epub 2024 May 22. PMID 38782232
- [Derived] Li Y, Wong A, Chung WM, Li M, Molasiotis A, Bressington D, Ma CZ, Kor PPK, Yeung WF. Evaluation of a Physical-Psychological Integrative (PPI) intervention for community-dwelling spinal cord injury survivors: Study protocol of a preliminary randomized controlled trial. PLoS One. 2023 Mar 20;18(3):e0282846. doi: 10.1371/journal.pone.0282846. eCollection 2023. PMID 36940214